CLINICAL TRIAL: NCT02122900
Title: Assessment of the Role of Balloon Aortic Valvuloplasty in the Management of Patients With Aortic Stenosis
Brief Title: Prospective Balloon Aortic Valvuloplasty
Acronym: BAV
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 013-142
Record Dates: First submitted 2014-03-03; First posted 2014-04-25 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary objective of this study is to determine the reasons for balloon aortic valvuloplasty (BAV) in the current clinical setting and to determine the outcomes of BAV in patients with aortic stenosis. The ultimate aim is to establish the safety, effectiveness, and appropriate role of BAV therapy as definitive therapy (palliation) or as a "bridge" to surgical aortic valve replacement (SAVR) or transcatheter aortic valve replacement (TAVR).

DETAILED DESCRIPTION:
Study Objectives:

1. To assess the volume of BAV procedures and success of the procedure as a 'bridge' to AVR/TAVR (percent of BAV patients that go on to receive valve replacement).
2. To establish the demographic profile of the patients having a BAV with clear determination of the primary indication for the BAV.
3. To collect baseline, 30-day, 3 and 6 month, and 1 year patient data to assess improvement in primary cardiac condition (AVA, EF & GRAD) and other primary endpoint conditions and symptomology according to pre-operative BAV rationale (e.g., renal function, chronic obstructive pulmonary disease, etc - see inclusion criterion).
4. To assess patient Quality Of Life prior to procedure and at all follow-up time points through to 1-year post-procedure
5. To assess patient's Resilience at baseline and 30 day follow-up using the Connor-Davidson 10 Resilience Scale.
6. To assess post-operative rate of stroke and other complications (according to VARC2 definitions ).
7. To identify the survival in relation to the treatment indication for BAV.

Background:

BAV is a percutaneous treatment for severe aortic stenosis with a balloon catheter inside the valve. The balloon stretches the valve open, in an effort to increase the opening size of the valve and improve blood flow.

While the procedure offers relief from symptoms, the preferred alternative is aortic valve replacement. The Cardiology/American Heart Association (ACC/AHA) Guidelines on Valvular Heart Disease assert that BAV should be limited to serving as a bridge to surgery in those with compromised hemodynamic status or as a method for palliation of symptoms in those who are not candidates for AVR (Class IIb).

With the commercial release of the Edwards Sapien transcatheter aortic valve system and increasing availability of TAVR, patients previously bridged to inclusion in TAVR feasibility trials with BAV might proceed more directly to TAVR. Thus an important challenge will be to better define the relative role for TAVR and of palliative BAV, especially in extreme-risk patients for whom the survival benefit of successful TAVR may be limited due to other life-threatening comorbid conditions.

A retrospective chart review of patients that had undergone BAV from 2006 to May 2013 was performed. Several indications were identified in relation to this surgical intervention (palliative therapy from the outset; a means to 'bridge' a patient to operable status / treatment; therapy for patients under consideration for TAVR but delayed due to trial constraints; and as ultimate therapy because patients declined further treatment). Unfortunately, however, patient category determinations were made post-hoc, and proved problematic to properly validate. The current study proposes to rectify that problem by collecting definitive diagnostic intention prior to study inclusion.

Methods of Proposed Research:

The study is a prospective collection of patient indication, procedural, and intermediate outcomes for all patients undergoing BAV. Data from hospital records, 30-day, 3 month, 6 month, and 1-year follow-up clinic visits and all other subsequent clinic and hospital records through to 1-year post-procedure will be collected.

Study Design:

With a minimum enrollment of 100 total patients, the estimated time period of this study is 6 months + 1 year for all baseline and follow-up data collection (beginning 6/2013 through 10/2014). This estimate is based on an average monthly rate of 7 BAV procedures at Medical City, and 10 at the Heart Hospital Baylor Plano.

Schedule of Assessments/Data Collection:

Pre-procedure: Kansas City QOL and Connor-Davidson 10 Resilience Scale will be assessed pre-procedure gained from all consenting patients prior to BAV. Indication for BAV will be obtained by a case report form for all patients.

Hospitalization period: All other data will be collected from existing medical records for hospitalization and for BAV procedure through to discharge, as well as all inpatient hospital visits following BAV through to 1 year follow-up.

30 day, 3 month, 6 month and 1 year clinic follow-up: Clinic follow-up will re-assess parameters of cardiac function, as well as pulmonary, and/or renal function as deemed necessary for evaluation of procedural "success" based on pre-BAV indicators. Telephone follow-up will be performed for any patients that fail to appear for clinic visits. QOL from all patients who have consented to QOL assessment will be obtained at each time point. The Connor-Davison 10 Resilience Scale will be collected at the 30 day follow-up visit.

Statistical & Analytical Methods:

The endpoint variables are procedural mortality, survival post intervention and other major adverse event (the following clinical endpoints will be queried as per VARC2 recommendations: mortality, stroke, myocardial infarction, bleeding complications, acute kidney injury, vascular complications, conduction disturbances and arrhythmias, and other relevant complications not previously categorized).

Indication for BAV will be the primary planned comparison, with additional analyses planned for demographic factors (age, gender, race/ethnicity, height, weight, and BMI, and body surface area (BSA). Changes in cardiac function (output in l/min, ejection fraction, aortic peak velocity in m/s, aortic valve area in cm2, aortic valve gradient in mmHg) will be compared in all patients with echocardiography. Definition of success will also assess change in renal function (lab creatinine values), and pulmonary (Fev1/DLCO) values, and pre-post score QOL and resilience scale changes.

Procedural variables will include balloon specifications, number of balloons used for each patient, number of times each balloon has been dilated, and complications. The latter will be distinguished in procedural and post procedural adverse events.

The results will be shown as mean and standard deviation, proportion of patients of the total numbers who had a BAV. The cardiac catheter lab parameters before and after the BAV procedure will be contrasted using a student's paired both tail T-Tests. A p value of less than 0.05 will be considered significant. Categorical variables will be compared using a chi- square test. The association between the risk factors and the outcome of interest will be tested with a Cox proportional hazards model. In addition Kaplan-Meier survival curves will be used to determine the time from BAV to procedural death and overall survival differentiated by each type of BAV indication.

Data Monitoring:

All data will be reviewed by Data Advisory Group for completeness and accuracy.

ELIGIBILITY:
Inclusion criteria:

Patients will be identified in the valve clinics and from the cath lab schedules. All patients who are scheduled to have a BAV during the study period in the cath lab at MCD and THHBP for whom a definitive pre-procedure BAV indication including the following will be eligible for enrollment:

* BAV as palliation
* BAV offered as a means of assessment for a change to operable status (a 'bridge' to decision). Patients in this category will be classified by the procedure physician as to the primary reason of 'bridge' decision - these reasons would include:

  * Diagnostic
  * Shortness of Breath- Aortic stenosis vs. other etiology such as COPD
  * Lack of Energy- Aortic stenosis vs. other etiology
  * LV Dysfunction - Aortic stenosis vs. cardiomyopathy
  * Therapeutic- determination of improvement to receive treatment
  * Frailty - Factors: grip strength, 5 meter walk time, Katz Index of Independence in Activities of Daily Living (Katz ADL), serum Albumin
  * Immobility - Reason for immobility and current assistive device will be documented
  * Stage IV chronic kidney disease - Cockoft- Gault formula (GRF 15-29 mL/min/1.73 m2) or high procedural risk for progression to dialysis dependence
  * End stage renal disease currently on dialysis Acute kidney Injury - (Varc 2)
  * Severe left ventricular dysfunction - BAV to improve EF (VARC 2) LVEF < 35% without contractile reserve
  * NYHA class IV congestive heart failure
  * Active bleeding
  * Urgent or emergent clinical status
  * Severe liver disease (VARC 2)
  * Active Infection
  * Other cause:_______________________________

The Kansas City Cardiomyopathy questionnaire (KCCQ), a quality of life (QOL) assessment, and the Connor-Davidson 10 Resilience Scale will be collected from all patients for whom informed consent is obtained by the study coordinators to administer the QOL assessment and resilience scale.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Aortic Stenosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
BAV outcome as a successful "bridge to TAVR/AVR" procedure. | Up to 1 year post BAV.
  This is an observational study intended to collect re-world safety outcomes of BAV and delineate if patients that undergo this procedure to improve their clinical status actually improve to a point that they qualify for a definitive treatment for their aortic stenosis.

SECONDARY OUTCOMES:
Measurement of improvement in primary cardiac function and symptomatology. | Up to 1 year post BAV.
  This is an observational study intended to collect re-world safety outcomes of BAV and delineate if patients that undergo this procedure to improve their clinical status actually improve to a point that they qualify for a definitive treatment for their aortic stenosis. Patients that undergo BAV will be followed up to 1 year post-BAV with NYHA class, quality of life scores and cardiac function (utilizing echocardiography) being tracked.

CONTACTS AND LOCATIONS:
Overall Officials: Molly Szerlip, MD, Principal Investigator — Baylor Research Instute
Locations (2):
- United States (2):
  - Medical City, Dallas, Texas
  - The Heart Hospital Baylor, Plano, Texas